CLINICAL TRIAL: NCT06931639
Title: Suicide Preventive Psychosocial Treatment for Youths: A Randomized Controlled Trial
Brief Title: Suicide Preventive Psychosocial Treatment for Youths
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Johan Bjureberg, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAFETYRCT2025; 2024-00196 (Other Grant/Funding Number: Swedish Research Council)
Record Dates: First submitted 2025-04-07; First posted 2025-04-17 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Suicide Attempt; Suicidal and Self-injurious Behavior; Suicide Attempted; Suicide, Attempted
Keywords: Safe Alternatives for Teens and Youths; Self-injurious Behavior; Suicide Attempt; Suicidal Behavior
MeSH Terms: conditions — Suicide, Attempted; Self-Injurious Behavior | interventions — Safety

STUDY DESIGN:
Intervention Model Description: Single-blind parallel-group randomized controlled multisite trial
Who Masked: Outcomes Assessor
Masking Description: Participants will be informed that they will be allocated to one of two psychosocial interventions addressing suicidality. Participants cannot be completely blinded; however, information about the two interventions will be kept to a minimum in the informed consent to avoid nocebo. Therapists who recruit participants and outcomes assessors will be blinded to the randomization sequence, and outcomes assessors will also be blinded to time-point. All participants will receive instructions not to reveal their treatment condition to the outcomes assessor. To assess the integrity of the blinded ratings, the blinded assessors will be instructed to record if the family accidentally revealed the condition, guess the participant's treatment allocation and motivation for their guess. If an assessor becomes unblinded, subsequent assessments for that participant will be conducted by a different assessor. Blinding will be broken after FU3 but masked assessors will remain blinded through follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safe Alternatives for Teens and Youth (SAFETY) (Experimental): SAFETY is a transdiagnostic cognitive-behavioral family treatment informed by Dialectical Behavior Therapy (DBT) and Multisystemic Therapy (MST). The twelve week long treatment is principle based, structured in phases, and individually tailored based on a cognitive-behavioral fit analysis that specifies key risk and protective processes. Each session contains one individual component for youth and parents respectively, and one family component where youth and parents work together with therapists to practice skills identified as critical for preventing future suicidal behavior. Treatment targets are arranged in a SAFETY Pyramid, consisting of (a) safe settings; (b) safe people; (c) safe activities and actions; (d) safe thought; and (e) safe stress reactions, emphasizing strengthening protective support and validation within the family and/or social environment surrounding the youth.
  Interventions: Behavioral: Safe Alternatives for Teens and Youth (SAFETY)
- Enhanced Treatment As Usual (Active Comparator): Enhanced Treatment As Usual (ETAU) consists of treatment as usual delivered by community clinicians enhanced by the evidence-informed Stanley-Brown Safety Planning Intervention, adapted for adolescents (e.g. involving both youth and parents) and to a Swedish context by the Swedish Association for Child and Adolescent Psychiatry and supervised by the research group. The adapted Safety Planning intervention include an assessment of current and future risk and protective factors for suicide, current and future suicide risk, and an individualized safety plan. We will ensure that the control intervention Safety Planning is delivered in a safe and comparable way across regions. Patients in both conditions will have access to standard care (including pharmaceutical treatment), as well as inpatient care as deemed necessary. The level of standard care will be carefully measured throughout the trial and included in statistical sensitivity analyses.
  Interventions: Behavioral: Enhanced Treatment As Usual

INTERVENTIONS:
Behavioral: Safe Alternatives for Teens and Youth (SAFETY) — Please see description of experimental arm (arm one)
  Arms: Safe Alternatives for Teens and Youth (SAFETY)
Behavioral: Enhanced Treatment As Usual — Please see description of active comparator arm (arm two).
  Arms: Enhanced Treatment As Usual

SUMMARY:
Suicide is the leading cause of death amongst 10-18-year-olds in Sweden. Suicide attempts are the strongest predictor of subsequent death by suicide, often lead to inpatient care, and are associated with substantial societal costs, making suicide attempts a critical target in psychiatric intervention research. Although youths attempting suicide are typically assessed and treated for potential comorbid psychiatric conditions, there is currently no trans-diagnostic evidence-based treatment specifically targeting suicidal behavior. To fill this gap, the Safe Alternatives for Teens and Youths (SAFETY) was developed. SAFETY is a transdiagnostic family-based cognitive-behavioral suicide prevention program that has shown promise but more studies are needed.

The overall objective of this project is to evaluate the efficacy, durability, and cost-effectiveness of the SAFETY intervention, a scalable suicide prevention intervention that can be offered immediately following a youth suicide attempt, in a fully powered single-blind randomized controlled superiority trial. Our primary hypothesis is that the SAFETY intervention will be superior to Enhanced Treatment As Usual (enhanced with the evidence-based intervention safety planning) in reducing the proportion of suicide reattempts. Moreover, we predict that these improvements will be maintained for up to 60 months post-treatment. Finally, we expect that SAFETY will be cost-effective compared to the control intervention, both at the primary endpoint and in the longer term.

DETAILED DESCRIPTION:
The overall objective of this project is to evaluate the efficacy, durability, and cost-effectiveness of the SAFETY intervention, a scalable suicide prevention intervention that can be offered immediately following a youth suicide attempt, in a single-blind randomized controlled multisite superiority trial.

PRIMARY OBJECTIVE To determine the clinical efficacy of SAFETY for reducing suicide re-attempt (as measured by the masked assessor-administered C-SSRS) in youths with a recent suicide attempt, compared with enhanced treatment as usual within child and adolescent mental health care (E-TAU). The primary endpoint is the follow-up 3 months post-treatment.

SECONDARY OBJECTIVES

1. To determine the clinical efficacy of SAFETY for nonsuicidal self-injury, global functioning, anxiety, depression, and hopelessness in youths with a recent suicide attempt, compared with E-TAU. The primary endpoint is the follow-up 3 months post-treatment.
2. To evaluate the clinical efficacy of SAFETY for a composite outcome of suicide attempts and nonsuicidal self-injury, in order to enable comparison with other studies.
3. To establish the 12-month durability of the treatment effects.
4. To conduct a health-economic evaluation of SAFETY for youth with a recent suicide attempt, compared with E-TAU, from multiple perspectives, both in the short term (primary endpoint) and the long term (12-month follow-up).
5. To test predictors and moderators of treatment effect, including factors related to baseline levels of the outcomes, comorbidity, personality, family functioning, parental factors, school experience, peer support, and traumatic experiences.
6. Test whether emotion regulation, thwarted belongingness and perceived burdensomeness, parental invalidation, and family functioning mediate treatment outcome.
7. Long-term follow-up from post-treatment to 60-month post-treatment including patient-reports and parent-reports, as well as psychiatric disorders, clinical care consumption, pharmacological prescriptions, employment status, and academic performance retrieved from registries.

ELIGIBILITY:
Inclusions criteria:

1. Suicide attempt in the last 3 months
2. Age 10-17 years
3. At least one primary caregiver (multiple is allowed) willing to participate in treatment

Exclusion criteria:

1. Symptoms obstructing participation in assessments or treatment
2. Insufficient understanding of the Swedish language in youth and/or caregiver
3. Enrolled in Dialectical Behavioral Therapy

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 282 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Suicide Attempt Score of the Columbia Suicide Severity Rating Scale (C-SSRS) | Pre-treatment, immediately post-treatment, as well as 3-, 12-, 24- and 60-month post-treatment.
  The C-SSRS is a 22-item structured clinical interview assessing the frequency and severity of suicidal ideation, suicidal behaviors, and self-harm.

SECONDARY OUTCOMES:
Deliberate Self-Harm Inventory - Youth version (DSHI-Y). | Pre-treatment, immediately post-treatment, as well as 3-, 12-, 24- and 60-month post-treatment.
  The DSHI-Y used in this trial is a 8-item clinican-rated interview that will be used to assess presence and frequency (0 to ∞) of non-suicidal self-injury, where a higher score indicates higher frequency of non-suicidal self-injury. One item measuring non-suicidal intoxications has been added to the original DSHI-Y. The DSHI-Y is adapted for adolescents from the DSHI an empirically supported measure of various aspects of NSSI originally developed for use with adults. The DSHI has demonstrated good test-retest reliability and adequate concurrent validity among adolescents.
Work and Social Adjustment Scale, youth version (WSAS-Y) | Pre-treatment, immediately post-treatment, as well as 3-, 12-, 24- and 60-month post-treatment.
  WSAS-Y is a clinician-rated scale of impaired functioning in school, everyday life, friends and social life, recreation and hobbies and family and close relationships. The scale generates a global score ranging from 0 to 40, with higher scores indicating greater impairment.
Children's global assessment scale (CGAS) | Pre-treatment, immediately post-treatment, as well as 3-, 12-, 24- and 60-month post-treatment.
  The CGAS is a clinician rated single item 1-100 scale that integrates psychological, social, and academic functioning in children as a measure of psychiatric disturbance. Higher values represent better functioning.
Revised Children's Anxiety and Depression Scale, 25 item version (RCADS-25) | Pre-treatment, immediately post-treatment, as well as 3-, 12-, 24- and 60-month post-treatment.
  The RCADS-25, a shortened version of the Spence Child Anxiety Scale, is a child self-report measure of anxiety- and depression-related psychopathology, with six subscales; separation anxiety, social anxiety, generalized anxiety, panic disorder, obsessive-compulsive disorder and major depressive disorder, as well as a total anxiety-scale. Total range is 0-45, Likert scale ranging from 0-3, with higher values representing a worse outcome.
Beck's Hopelessness Scale (BHS) | Pre-treatment, immediately post-treatment, as well as 3-, 12-, 24- and 60-month post-treatment.
  Beck's Hopelessness Scale is a youth self-rated measure of hopelessness, with 20 dichotomous "true/false" items measuring hopelessness in three domains; feelings about the future, loss of motivation and expectations. A higher score indicates greater difficulties related to hopelessness.
Child Health Utility 9D (CHU-9D) | Pre-treatment, immediately post-treatment, as well as 3-, 12-, 24- and 60-month post-treatment.
  The CHU-9D is a youth-rated measure of health related quality of life for youth, with 9 items on a Likert scale ranging from 0-4. Scores range from 0-36, with a lower score indicating greater health-related quality of life.
Recovering Quality of Life (ReQoL) | Pre-treatment, immediately post-treatment, as well as 3-, 12-, 24- and 60-month post-treatment.
  Recovering Quality of Life is a parent-rated measure of health-related quality of life for adults, with 10 items on a Likert scale of 0-4, yielding a range of 0-40, where a higher score indicate higher quality of life.
Trimbos/iMTA questionnaire for Costs associated with Psychiatric illness (TIC-P) | Pre-treatment, immediately post-treatment, as well as 3-, 12-, 24- and 60-month post-treatment.
  The TIC-P is a 37-item measure assessing healthcare and societal resource use, including for example items on healthcare resource use, medications, school absenteeism, and parental productivity loss. Rated by parents.

OTHER OUTCOMES:
Self-harm | Pre-treatment, immediately post-treatment, as well as 3-, 12-, 24- and 60-month post-treatment.
  Composite outcome of suicide attempts (C-SSRS) and nonsuicidal self-injury (DSHI-Y) ranging from (0 to ∞), in order to enable comparison with other studies.
Borderline Personality Feature Scale for Children-11 (BPFS-C-11) | Pre-treatment
  The BPFS-C-11 is a youth-rated 11-item measure of borderline personality features for children 9 - 18 years old. The BPFS-C-11 includes indicators of borderline pathology such as affective instability, identity problems, and negative relationships. Item responses are on a 5-point Likert scale, yielding a range of 11-55, with higher scores indicating higher levels of borderline features.
Levels of Personality Functioning Questionnaire 12-18 (LoPF-Q 12-18) | Pre-treatment
  LoPF-Q 12-18 is a youth-rated 20-item measure rated on a scale of 0-4, yielding a range of 0-80, where a higher score indicates higher impairment in personality functioning. LoPF-Q is developed for use in adolescent populations between 12 and 18 years to assess the dimensions of personality functioning: identity, self-direction, empathy, and intimacy.
Borderline Symptom List Supplement (BSL-Supplement) | Pre-treatment, immediately post-treatment, as well as 3-, 12-, 24- and 60-month post-treatment.
  The BSL-Supplement is a youth-rated 9-item measure of self-destructive behaviors under the past 7 days, with answers ranging from "Not at all" to "Daily or even more often". Higher scores indicate a higher frequency of self-destructive behaviors.
Credibility/Expectancy Questionnaire (CEQ) | Two weeks after treatment initiation.
  CEQ is a youth and parent-rated 6-item measure of treatment credibility and expectancy. Scale points range from 0-9, and 0-100%, where higher scores indicate greater credibility and expectancy.
Adverse events | Immediately post-treatment
  Participants (parents and youths) are asked to report and rate the discomfort of the eventual adverse events caused by their participation in the treatment. Adverse events are also continuously screened for, recorded, and monitored by study personnel.
Credibility/Expectancy Questionnaire, short (CEQ) | Pre-treatment
  At baseline, we use one item from the CEQ addressing treatment expectancy. Scale points for this item range from 0-100%, where a higher score indicates higher expectancy. This item is both youth and parent-rated.
Client Satisfaction Questionnaire (CSQ) | Immediately post-treatment
  The CSQ is a youth- and parent-rated 8-item measure on a 4-point scale measuring different aspects of satisfaction with treatment, e.g., perception of quality of treatment, if the treatment adequately addressed their needs and overall satisfaction. The score ranges from 8-32, where a higher score indicates higher treatment satisfaction.
Difficulties in Emotion Regulation Scale, Short form (DERS-16) | Pre-treatment, immediately post-treatment, as well as 3-, 12-, 24- and 60-month post-treatment
  The DERS-16 is a youth- and parent-rated measure of difficulties in emotion regulation, with 16 items rated on a 1-5 Likert scale, with scores ranging from 16-80 and higher scores indicating greater difficulties in emotion regulation.
Cognitive Emotion Regulation Questionnaire (CERQ, Self-blame sub-scale) | Pre-treatment, immediately post-treatment, as well as 3-, 12-, 24- and 60-month post-treatment
  The CERQ is a youth-rated measure of cognitive emotion regulation. The self-blame sub-scale contains 4 items on a Likert scale ranging from 1-5. Scores range from 4-20, and higher scores indicate greater difficulties with self-blame.
Behavioral Emotion Regulation Questionnaire (BERQ, Seeking Social Support and Actively Approaching sub-scales) | Pre-treatment, immediately post-treatment, as well as 3-, 12-, 24- and 60-month post-treatment
  The BERQ is a youth-rated measure of behavioral emotion regulation. The sub-scales Seeking Social Support and Actively Approaching contains 8 items on a Likert scale ranging from 1-5. Scores range from 8-40. A higher score indicates greater behavioral emotion regulation regarding seeking social support and actively approaching.
Interpersonal Needs Questionnaire (INQ) | Pre-treatment, immediately post-treatment, as well as 3-, 12-, 24- and 60-month post-treatment
  The INQ is a youth-rated measure containing 15 questions rated on a Likert scale of 1-7. The INQ measures beliefs about the extent to which individuals believe their need to belong is met or unmet, as well as the extent to which they perceive themselves to be a burden on the people in their lives. Scores range from 15-105, with higher scores indicating worse outcomes.
Family Assessment Device (FAD, General Functioning sub-scale) | Pre-treatment, immediately post-treatment, as well as 3-, 12-, 24- and 60-month post-treatment
  The FAD is a 60-item questionnaire that measures an individual's perceptions of his/her family, rated by youth and parents. We utilize a subset of 6 questions from the General Functioning Scale of the FAD. Scores range from 0-18, with higher scores indicating greater general family functioning.
Hierarchical Personality Inventory for Children-30 (HiPIC-C-30, Neuroticism and Conscientiousness subscales) | Pre-treatment
  HiPIC-C-30 is a 30-item measure (Likert scale 1-5) assessing the personality constructs of neuroticism, extraversion, openness, conscientiousness, and agreeableness. We will use the subscales measuring neuroticism and conscientiousness, resulting in a 12-item measure, rated by youths and parents. Scores range from 6-30 within each subscale, and higher scores indicate more neuroticism and conscientiousness, respectively.
Child Trauma Screen (CTS) | Pre-treatment
  The CTS is a youth-rated 10-item screening measure of trauma exposure and PTSD symptoms for children ages 6-17. Six questions related to reaction/PTSD symptoms are summed to create a reaction score (rated on a Likert scale of 0-3) yielding a range of 0-18, where a cutoff score of 6 or greater indicates a high likelihood of PTSD diagnosis.
Functioning | Pre-treatment, immediately post-treatment, as well as 3-, 12-, 24- and 60-month post-treatment.
  Three self-composed youth-rated questions measuring school functioning, functioning with peers and family functioning. Each question is rated separately and on a Likert scale from 0-11, with a higher score indicating greater functioning in each respective functioning domain.
School Success Profile (SSP, Parental Encouragement sub-scale) | Pre-treatment, immediately post-treatment, as well as 3-, 12-, 24- and 60-month post-treatment.
  Subscales from the SSP will be rated by youths and parents, respectively. Youth will answer 12 questions relating to parental and peer support as well as attitudes toward school. Parents will answer 4 questions relating to parental support. Responses are rated on a 0-4 Likert scale. Higher scores indicate greater support and positive attitudes.
Coping with Children's Negative Emotions Scale Adolescent version(CCNES-A) | Pre-treatment, immediately post-treatment, as well as 3-, 12-, 24- and 60-month post-treatment.
  The CCNES-A is a measure of parental coping responses in response to youths' negative emotions. The CCNES-A version used in this study consists of nine hypothetical scenarios, accompanied by six theoretically meaningful types of responses (including how well the parent handles their own emotions triggered by the hypothetical situation with the youth) rated by the youth as well as the parent on a Likert scale ranging from 1-7. Higher scores in each subscale representing a response style indicate a higher tendency of the response style.
Parenting Distress Index - Short (PDI-Short) | Pre-treatment, immediately post-treatment, as well as 3-, 12-, 24- and 60-month post-treatment.
  The PDI-short is parent-rated and includes 2 questions about parenting distress (rated on a Likert scale of 1-5), where higher scores indicate more stress.
Parental Abuse Scale (PAS) | Pre-treatment, immediately post-treatment, as well as 3-, 12-, 24- and 60-month post-treatment.
  The PAS is youth-rated and contains 7 questions on a Likert scale from 0-4 assessing how often aversive parental behaviors have been experienced by the youth. Scores range from 0-28 and higher scores indicate more frequent experiences of aversive parental behaviors.
Register-based outcomes | 24- and 60-month post-treatment
  Data on psychiatric disorders, clinical care consumption, pharmacological prescriptions, employment status, and academic performance will be derived from national population-based registers.
Parent Self-Efficacy for Suicide Scale | Pre-treatment, immediately post-treatment, as well as 3-, 12-, 24- and 60-month post-treatment.
  The Parent Self-Efficacy for Suicide Scale is a parent-rated measure of self-efﬁcacy, or conﬁdence, regarding parents' ability to engage in nine activities to prevent or assist their child in managing a suicidal crisis, and parent expectations of adolescents' risk of subsequent suicide. The measure contains 12 items, rated on a scale of 0 (not at all conﬁdent) to 10 (completely conﬁdent), with an anchor of 5 (somewhat conﬁdent), resulting in a range of 0-120. The measure includes two subscales: self-efficacy (9 items) and expectation (3 items). Higher scores indicate higher levels of self-efficacy, and greater expectations of a positive outcome regarding suicidality.
Patient Health Questionnaire (PHQ-9) | Pre-treatment, immediately post-treatment, as well as 3-, 12-, 24- and 60-months post-treatment.
  The PHQ-9 is a parent-rated measure used for screening, diagnosing, monitoring and measuring the severity of depression. The measure contains 9 items, rated on a scale of 0 to 3, resulting in a range of 0-27, where a higher score indicates higher levels of depression.

CONTACTS AND LOCATIONS:
Locations (5):
- Sweden (5):
  - Child and Adolescent Mental Health Services, Region Skåne, Helsingborg
  - Child and Adolescent Psychiatry, Region Värmland, Karlstad
  - Child and Adolescent Mental Health Services, Region Halland, Kungsbacka
  - Child and Adolescent Mental Health Services, Region Stockholm, Stockholm
  - Child and Adolescent Psychiatry, Region Uppsala, Uppsala

IPD SHARING:
Plan to Share IPD: No
Patient-level data are not publicly available due to national (Swedish) and EU legislation but could be made available from the corresponding author upon reasonable request following approval from the Swedish Ethical Review Authority.